CLINICAL TRIAL: NCT07224347
Title: Aspirin in Reducing Events in the Elderly-Extension (ASPREE-XT)
Status: Active, not recruiting | Type: Observational
Sponsor: Anne Murray (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Bayer (Industry); Monash University (Other); Berman Center for Outcomes and Clinical Research (Other); National Institute on Aging (NIA) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Anne Murray, Principal Investigator, Staff Endocrinologist, Hennepin Healthcare Research Institute
Organization: Hennepin Healthcare Research Institute (Other)
Other Study IDs: 201904807; U19AG062682 (NIH)
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-01

CONDITIONS: Functional Disability; Dementia; Heart Disease; Stroke; Cancer; Bleeding; Depression; Frailty
Keywords: Aspirin; Prevention; Healthy; Over 70 years old; ASPREE; Aspirin in Reducing Events in the Elderly; Australia; Functional Disability; Dementia; Heart Disease/ Stroke; Cancer; Bleeding; Frailty; Community-Dwelling; Older Adult
MeSH Terms: conditions — Dementia; Heart Diseases; Stroke; Neoplasms; Hemorrhage; Depression; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aspirin: 100 mg enteric-coated aspirin
- Placebo: Placebo

SUMMARY:
ASPREE-XT is a post-treatment, longitudinal observational follow-up study of ASPREE participants. Although the ASPREE trial medication was ceased, the study activity was not stopped and ASPREE participants are continuing with scheduled visits and phone calls. An observational follow-up phase (ASPREE-XT), began in January, 2018. This will enable the monitoring of possible delayed effects of aspirin treatment, primarily on cancer incidence, metastases and mortality. In addition to monitoring the incidence of malignancy within the ASPREE cohort, the opportunity will be taken to observe any other residual effects of aspirin on the endpoints being monitored in the cohort. Continuity of contact with study participants is the key to retention of the cohort for any ongoing or future studies.

DETAILED DESCRIPTION:
ASPREE-XT is a longitudinal, observational follow-on study of ASPREE participants.

The methodology of ASPREE-XT is based closely on ASPREE [ASPREE investigator group, 2013; www.aspree.org; McNeil et al. 2017]. Clinical, neurocognitive and physical function measurements, questionnaires for mood, quality of life, physical ability and collection of personal health, demographic and lifestyle details are the same in ASPREE-XT as those conducted and described for ASPREE.

Since ASPREE-XT is an observational study, the endpoints for ASPREE will be collected and adjudicated in a similar way for ASPREE-XT but will be referred to as ASPREE-XT Outcomes. These will not be divided into primary and secondary endpoints.

In 2018, participants were invited to enroll in ASPREE-XT. At the first ASPREE-XT study visit, or via mail, they were provided with an information sheet and consent form for the study Participants who wish to only be contacted by phone were provided with information and a consent form by mail with health and other study data collected by phone call.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* African American and Hispanic persons age 65 or older
* Any person from another ethnic minority group and Caucasian persons age 70 or older
* Willing and able to provide informed consent, and willing to accept the study requirements

Exclusion Criteria:

* A history of a diagnosed cardiovascular event
* A serious intercurrent illness likely to cause death within the next 5 years, such as terminal cancer or obstructive airways disease
* A current or recurrent condition with a high risk of major bleeding, ex: cerebral aneurysm
* Anemia
* Absolute contraindication or allergy to aspirin
* Current participation in a clinical trial
* Current continuous use of aspirin or other anti-platelet drug or anticoagulant for secondary prevention. People with previous use of aspirin for primary prevention may enter the trial, provided they agree to cease existing use of aspirin and understand that they may be subsequently randomly allocated to low dose aspirin or placebo.
* A systolic blood pressure ≥180 mmHg and / or a diastolic blood pressure ≥105 mmHg
* A history of dementia
* Severe difficulty or an inability to perform any one of the 6 Katz ADLs
* Non-compliance to taking pill

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Study Population: Men and women recruited from the United States and Australia.
  * African American and Hispanic persons age 65 or older in the U.S.
  * Any person from another ethnic minority group and Caucasian persons age 70 or older
  * Willing and able to provide informed consent, and willing to accept the study requirements
Sampling Method: Probability Sample
Enrollment: 19114 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Death from any cause or incident dementia or permanent physical disability. | Planned 5-year time frame
  These categories of disability are defined, respectively, as a) all-cause mortality, b) the assessment of dementia by DSM-IV criteria or c) the onset of 'a lot of difficulty' or 'inability' to perform independently, any one of 6 Katz ADLs.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Murray, MD, MSc, Principal Investigator — Berman Center for Outcomes and Clinical Research; John McNeil, MBBS, PHD, Principal Investigator — Monash University
Locations (36):
- United States (22):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Howard University, Washington D.C., District of Columbia
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory/ Atlanta VAMC, Atlanta, Georgia
  - Rush Alzheimer's Disease Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - LSU Health Sciences- Shreveport, Shreveport, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - HealthPartners Research Institute, Minneapolis, Minnesota
  - Phalen Village Clinic, Saint Paul, Minnesota
  - Wake Forest University Baptist Medical Center, Greensboro, North Carolina
  - The Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Health Sciences Research Center, Pittsburgh, Pennsylvania
  - Kent County Memorial Hospital, Pawtucket, Rhode Island
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Regional Academic Health Center, Harlingen, Texas
  - UT Health Science Center at San Antonio, San Antonio, Texas
- Australia (14):
  - Clinical Trials Unit, The Canberra Hospital, Garran, Australian Capital Territory
  - Illawarra Health and Medical Research Institute, University of Wollongong, Wollongong, New South Wales
  - Discipline of General Practice, School of Population Health, University of Adelaide, Adelaide, South Australia
  - Greater Green Triangle University, Mount Gambier, South Australia
  - University of Tasmania Rural Clinical School, Burnie, Tasmania
  - The Menzies Institute for Medical Research, University of Tasmania, Hobart, Tasmania
  - University of Tasmania Newnham Campus, Launceston, Tasmania
  - Bendigo Regional Clinical School, Bendigo, Victoria
  - Geelong Hospital, Geelong, Victoria
  - Monash Mildura Regional Clinical School, Mildura, Victoria
  - University of Ballarat, Mount Helen, Victoria
  - Monash Gippsland Regional Clinical School, Traralgon, Victoria
  - The South West Alliance of Rural Health (SWARH), Warrnambool, Victoria
  - Gateway Community Health, Wodonga, Victoria